CLINICAL TRIAL: NCT02087917
Title: A 4-week, Randomized, Placebo-Controlled, Double-Blind, Efficacy and Safety Study of HS-25 in Adults With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-25-III
Record Dates: First submitted 2014-03-05; First posted 2014-03-14 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Primary Hypercholesterolemia
Keywords: hypercholesterolemia; cholesterol absorption inhibitor; placebo-controlled trial
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- HS-25 5 MG (Active Comparator)
  Interventions: Drug: HS-25
- HS-25 10 MG (Active Comparator)
  Interventions: Drug: HS-25
- HS-25 20 MG (Active Comparator)
  Interventions: Drug: HS-25
- HS-25 30 MG (Active Comparator)
  Interventions: Drug: HS-25

INTERVENTIONS:
Drug: HS-25 — Assigned study drug (HS-25 or placebo) is to be administered orally once daily in the morning with or without food. Treatment duration 4 weeks.
  Arms: HS-25 10 MG; HS-25 20 MG; HS-25 30 MG; HS-25 5 MG
Drug: Placebo — Assigned study drug (HS-25 or placebo) is to be administered orally once daily in the morning with or without food. Treatment duration 4 weeks.
  Arms: Placebo

SUMMARY:
To determine the efficacy of HS-25 (5, 10, 20 or 30 mg) in reducing low density lipoprotein-cholesterol (LDL-C) levels after a 4-week period of treatment in adults with primary hypercholesterolemia.

DETAILED DESCRIPTION:
This is a 4-week, randomized, double-blind, placebo-controlled study designed to assess the effects of the cholesterol absorption inhibitor HS-25 on LDL-C levels in adults who have untreated LDL-C levels ranging from 130-189 mg/dL and fasting triglyceride levels < 350 mg/dL. Eligibility is restricted to 18-65 year old men or women who are using a highly effective birth control method or are not of childbearing potential. Patients with diabetes, a history of myocardial infarction or other clinical evidence of atherosclerotic vascular disease are not eligible for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Men, or women using a highly effective birth control method or not of child-bearing potential, who are 18 to 65 years of age at Visit 1 (screening visit).
* LDL-C 130 to 189 mg/dL (inclusive) on a cholesterol lowering diet but no lipid modifying drug treatment for at least 6 weeks. A qualifying LDL-C value must be obtained at the beginning and end of the placebo run-in (Visit 2 and Visit 3) and the Visit 3 value must be within 15% of the value at Visit 2, higher or lower; the average of both qualifying values must be in the range of 130 to 189 mg/dL (inclusive) for inclusion in the study.
* TG ≤ 350 mg/dL on a cholesterol lowering diet but no lipid modifying drug treatment for at least 6 weeks and TG levels must be ≤ 350 mg/dL at both Visit 2 and Visit 3
* Compliance of 80% to 120% with assigned study drug regimen during a 2 week placebo run-in phase.

Exclusion Criteria:

* Women who are pregnant or breast feeding.
* History of stroke, myocardial infarction, unstable angina, heart failure or any arterial revascularization procedure (eg, carotid, coronary, aorta, peripheral arterial).
* History of diabetes or glycosylated hemoglobin (HbA1c) > 6.5.
* History of moderate to severe lactose intolerance (eg, unable to drink a glass of milk).
* History of hospitalization for treatment of a major psychiatric disorder.
* History of drug or alcohol abuse as defined by the Diagnostic and Statistical Manual (DSM-5) within the prior 12 months.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months prior to screening.
* Hospitalization for a duration > 24 hours for any reason within the prior 3 months that, in the opinion of the investigator, may affect adherence to study procedures.
* History of a positive test for human immunodeficiency virus, hepatitis B or hepatitis C.
* History of cancer with the exception of well-treated basal cell or squamous cell carcinoma of skin, or in-situ cervical carcinoma.
* Presence of any condition which, in the opinion of the investigator, is likely to compromise completion of this trial or not be in the best interest of the subject.
* History of intolerance to ezetimibe.
* Participation in a prior study of HS 25.
* Participation in a study of an investigational drug or device within the prior 3 months unless subject has documentation of placebo administration in a placebo-controlled drug treatment trial only.
* Treatment with a fibric acid derivative (eg, fenofibrate, gemfibrozil), probucol, warfarin, systemic corticosteroid, cyclosporine or other immunosuppressant agent within the prior 12 weeks.
* Anticipated need or frequent use of acetaminophen (> 2 gm/day, that is required > 4x/week).
* Vitamins, herbal and dietary supplements must be discontinued at screening unless subject has been on a long-term daily regimen and agrees to continue this regimen during the study.
* Alanine aminotransferase (ALT) > 1.0 × upper limit of normal (ULN) at Visit 1, Visit 2 or Visit 3.
* Aspartate aminotransferase (AST) > 1.0 × ULN at Visit 1, Visit 2 or Visit 3.
* Unexplained (not due to exercise or strenuous activity) creatinine kinase increase > 2 × ULN at Visit 1, Visit 2 or Visit 3.
* Estimated glomerular filtration rate (Modification of Diet in Renal Disease) < 60 mL/min/1.73m2 at Visit 1, Visit 2 or Visit 3.
* Thyroid stimulating hormone outside of the normal range.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical disease (eg, infectious disease) must not be enrolled.
* Any other laboratory abnormality considered by the investigator to be clinically significant.
* Any subject with an electrocardiogram (ECG) having a QTc interval ≥ 450 msec, or any other abnormality considered by the investigator to be clinically significant at the end of placebo run-in (Visit 3) should not be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C after 4 weeks of double-blind treatment | 4 weeks

SECONDARY OUTCOMES:
Percentage of participants with reported adverse events during a 4-week period of treatment as a measure of safety and tolerability of HS-25 | 4 weeks
Percent change from baseline in LDL-C after a 1 and 2-week period of double-blind treatment | 1- and 2-weeks
Percent change from baseline in apoprotein B, non-high density lipoprotein-cholesterol, total cholesterol, triglycerides, high density lipoprotein-cholesterol and apoprotein A1 levels after a 1, 2 and 4-week period of treatment | 1-, 2- and 4-week periods
Mean concentration of HS-25 dose and its major metabolite (HS-25-M1) during treatment with HS-25 5, 10, 20 or 30 mg. | 1-, 2- and 4-week
Correlation between trough HS-25 and HS-25-M1 levels and percent change in LDL-C, apoA1, apoB, non-HDL-C, TC, TG, and HDL-C during a 4-week period of HS-25 treatment. | 1-, 2- and 4-week

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Liao, PhD, Study Director — Zhejiang Hisun Pharmaceuticals Co., Ltd
Locations (27):
- United States (27):
  - Chandler, Arizona
  - Phoenix, Arizona
  - West Hills, California
  - Doral, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - South Miami, Florida
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Auburn, Maine
  - Bethesda, Maryland
  - Methuen, Massachusetts
  - Trenton, New Jersey
  - Rochester, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Penndel, Pennsylvania
  - Greensboro, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia